CLINICAL TRIAL: NCT03399630
Title: Injection of Autologous Adipose Tissue for Treatment of Osteoarthritis in the Knee: A Controlled, Double-Blinded Trial
Brief Title: Injection of Autologous Adipose Tissue for Treatment of Osteoarthritis in the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aestique Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATOA-01
Record Dates: First submitted 2017-10-11; First posted 2018-01-16 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteo Arthritis Knee; Autologous Adipose Tissue

STUDY DESIGN:
Intervention Model Description: Double blind parallel groups assignment
Who Masked: Participant, Care Provider
Masking Description: Patient and treating physician are both blinded, being that neither are aware of which knee received the autologous adipose tissue injection and which knee received the placebo lactated ringers injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection of Autologous Adipose Tissue (Active Comparator): Treatment knee receives injection of 1.5 cc's of adipose tissue mixed with 1.5 cc's of Lactated Ringers
  Interventions: Other: Injection of Autologous Adipose Tissue
- Injection of Lactated Ringers (Placebo Comparator): Placebo control group receives injection of 3 cc's of Lactated Ringers with no adipose tissue
  Interventions: Other: Injection of lactated ringers

INTERVENTIONS:
Other: Injection of Autologous Adipose Tissue — Injection of Autologous Adipose Tissue to study the safety and efficacy of treating osteoarthritis
  Arms: Injection of Autologous Adipose Tissue
Other: Injection of lactated ringers — Injection of placebo lactated ringers to compare against the injection of autologous adipose tissue.
  Arms: Injection of Lactated Ringers

SUMMARY:
Evaluating the safety and efficacy of a single injection of autologous adipose tissue for treatment of osteoarthritis of the knee.

DETAILED DESCRIPTION:
This clinical trial is a single site, double blinded, paired within groups, controlled clinical study to investigate the safety and efficacy in the use of adult autologous adipose tissue for the treatment of pain associated with joint OA. The hypothesis of this trial is that the treatment will be safe and the proposed clinical outcome measures of reduced pain resulting from the treatment of OA of the knee joint with autologous adipose tissue will be superior to a placebo control treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral K-L Grade II through Grade IV osteoarthritis as diagnosed by physician review of weight bearing X-ray or MRI excluding subjects whose knee pain is caused by, (i) diffuse edema, (ii) displaced meniscus tear, (iii) lesion greater than 1 cm in any direction, or (iv) osteochondritis dissecans.
2. Study Participants must be willing to voluntarily give written Informed Consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed.
3. Males and females 40-75 years old.
4. Participants will be in good health (ASA Class I-II) with a BMI < 35.
5. Continued pain in the knee despite conservative therapies for at least 6 months.
6. Participants must present with a bilateral knee pain scores ≥6 and ≤16 using the short-form WOMAC pain (A1 subscale, 20 total points).
7. Must speak, read and understand English.
8. Subjects must be reasonably able to return for multiple follow-up visits.

Exclusion Criteria:

1. Participants who have had surgery of either knee within 6 months prior to the screening visit.
2. Participants who have had a major injury to either knee within 12 months prior to enrolling in the study.
3. Participants who have had an injection in either knee in the prior 6 months, including corticosteroids, viscosupplementation or platelet rich plasma (PRP).
4. Participants who have gout, rheumatoid arthritis, lupus arthropathy, psoriatic arthritis, avascular necrosis, severe bone deformity, infection of the knee joint, fibromyalgia, pes anserine bursitis, or neurogenic or vascular claudication.
5. Participants who have symptomatic OA of the hips, spine, or ankle that would interfere with the evaluation of the treated knee.
6. Participants that are unwilling to stop taking prescription pain medication 7 days prior to any visit.
7. Participants that are allergic to lidocaine, epinephrine or valium
8. History of bleeding disorders, anticoagulation therapy that cannot be stopped 3 days prior to injection
9. Subjects that use any form of tobacco to include e-cigarettes more than once a week within the last 6 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Safety - Incidence of Treatment-Emergent Adverse Events | 6 months
  Subjects will be monitored for adverse events

SECONDARY OUTCOMES:
Efficacy - Change in Pain Scores on the WOMAC Scale at All Follow-Up Visits | 1 week, 6 weeks, 3 months, and 6 months
  Patient outcomes for pain will be recorded
Efficacy - Change in Function Scores on the WOMAC Scale at All Follow-Up Visits | 1 week, 6 weeks, 3 months, and 6 months
  Patient outcomes for function will be recorded
Efficacy - Change in Stiffness Scores on the WOMAC Scale at All Follow-Up Visits | 1 week, 6 weeks, 3 months, and 6 months
  Patient outcomes for stiffness will be recorded

OTHER OUTCOMES:
Efficacy - Change in Pain Scores on the VAS Scale at All Follow-Up Visits | 1 week, 6 weeks, 3 months, and 6 months
  Patient outcomes for pain will be recorded
Efficacy - Change in Function Scores on the VAS Scale at All Follow-Up Visits | 1 week, 6 weeks, 3 months, and 6 months
  Patient outcomes for function will be recorded
Efficacy - Change in Stiffness Scores on the VAS Scale at All Follow-Up Visits | 1 week, 6 weeks, 3 months, and 6 months
  Patient outcomes for stiffness will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Lazzaro, MD, Principal Investigator — Aestique Ambulatory Surgical Center
Locations (2):
- United States (2):
  - Aestique Ambulatory Surgical Center, Greensburg, Pennsylvania
  - DNA Advanced Pain Treatment, Greensburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No